CLINICAL TRIAL: NCT03177226
Title: Safety & Feasibility of Functional Electrical Stimulation for The Treatment of Premature Ejaculation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Virility Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: VM II-Rev-001
Record Dates: First submitted 2017-05-28; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional TENS stimulation (Experimental): Short stimulation to identifying Sensory Threshold and Motor Threshold, followed by continuous functional electrical stimulation, throughout the entire self-stimulation phase [from full erection to ejaculation]
  Interventions: Device: Functional TENS stimulation
- Non-stimulation treatment (Sham Comparator): Short stimulation to identifying Sensory Threshold and Motor Threshold, followed by continuous non-functional electrical stimulation, throughout the entire self-stimulation phase [from full erection to ejaculation]
  Interventions: Device: Non-Functional TENS stimulation

INTERVENTIONS:
Device: Functional TENS stimulation — A short continuous electrical stimulation, beginning at 0 mAmp and gradually increased by +0.5 mAmp every 2-10 sec to identifying Sensory Threshold (Is) and Motor Threshold (Imc), followed by continuous functional electrical stimulation, throughout the entire self-stimulation phase, equal to his Icm'
  Other Names: 1427970 TensMed S82
  Arms: Functional TENS stimulation
Device: Non-Functional TENS stimulation — A short continuous electrical stimulation, beginning at 0 mAmp and gradually increased by +0.5 mAmp every 2-10 sec to identifying Sensory Threshold (Is) and Motor Threshold (Imc), followed by continuous non-functional electrical stimulation, throughout the entire self-stimulation phase, equal to his Icm'
  Arms: Non-stimulation treatment

SUMMARY:
Prospective, non-randomized, controlled, single-center study, to evaluate the efficacy of applied nominal electrical stimulation parameters given to premature ejaculation (PE) patients in order to prolong the ejaculatory latency time which will eventually increase the quality of their sexual life.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Clinical history of premature ejaculation
* Familiar with self- stimulation
* Ability to follow study instructions and complete study assessment tools
* Washout period of two weeks

Exclusion Criteria:

* History of cardio-vascular disorders
* Any type of implanted pacemaker/defibrillator
* Hypertension
* Diabetes Mellitus
* Local dermatological disease
* Local skin irritation/ lesions
* Any neurological disorder
* Any psychiatric disease and/or any psychiatric medications
* Any neoplastic disease in the past two years

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Procedure day
  All Self reported safety events (e.g. discomfort, pain, local irritation, local heat, noticeable changes in urination or bowl activity or any other complaint)
Change in ejaculation latency time | Procedure day
  The difference between patient ejaculation latency time under perineal functional electrical stimulation during self-stimulation, and latency time during self-stimulation while no electrical stimulation is applied

SECONDARY OUTCOMES:
Incidence of post-treatment Adverse Events | 72 hours
  Post treatment safety evaluation completed by subjects (using safety questionnaire)

OTHER OUTCOMES:
Effects of applied electrical stimulation on Erection using Self Reported - User Questionnaire | Procedure day
  Self reported - user questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Gruenwald, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No